CLINICAL TRIAL: NCT01944267
Title: Apically Positioned Flap, Free Gingival Graft and Apically Positioned Flap With Collagen Matrix Around Dental Implants
Brief Title: Procedures for Improving the Mucosa Around Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 10893
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Keratinized Mucosa; Dental Implants
MeSH Terms: interventions — Mucograft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Apically positioned flap (Active Comparator): Standard TUSDM Periodontology Clinic procedures will be followed. Local anesthesia will be achieved. Center of implant fixtures will be located. Crestal incision thru the center of implant fixture will be made. Implant fixture will be uncovered and healing abutment/s will be inserted. Horizontal incision at approximately 0.5mm coronal to buccalmucogingival junction will be made 1 tooth mesial to 1 tooth distal to the treating area.
  No vertical incision will be made Gingiva coronal to horizontal incision will remain intact Partial thickness flap will be prepared and displaced apically approximately 7mm from the horizontal incision and secured with sutures.
  Prepared surgical area will be measured apico-coronally and mesio-distally.
  Interventions: Procedure: Apically positioned flap
- Free Gingival Graft (Active Comparator): Standard Clinic procedures followed. Local anesthesia achieved. Center of implant fixtures located. Crestal incision thru center of fixture will be made.
  Implant fixture uncovered and healing abutment/s inserted. Horizontal incision at approx 0.5mm coronal to buccalmucogingival junction will be made 1 tooth mesial to 1 tooth distal to the treating area.
  No vertical incision made. Gingiva coronal to horizontal incision remains intact.
  Partial thickness flap prepared and displaced apically approximately 7mm from horizontal incision; secured with sutures. Prepared recipient bed measured apico-coronally and mesio-distally. Masticatory mucosa from palate of treating side (Right or Left) harvested according to size measured from recipient bed with width of approximately 5mm at line of measurement. Harvested graft material will be transplanted on recipient bed, lined with initial horizontal incision line with sutures
  Interventions: Procedure: Free Gingival Graft
- Apically positioned flap with Mucograft (Active Comparator): Standard TUSDM Periodontology Clinic procedures followed. Local anesthesia achieved.
  Center of implant fixtures will be located. Crestal incision thru the center of implant fixture will be made. Implant fixture will be uncovered and healing abutment/s will be inserted. Horizontal incision at approximately 0.5mm coronal to buccalmucogingival junction will be made 1 tooth mesial to 1 tooth distal to the treating area.
  No vertical incision will be made. Gingiva coronal to horizontal incision will remain intact. Partial thickness flap will be prepared and displaced apically approximately 7mm from the horizontal incision and secured with sutures.
  Prepared recipient bed will be measured apico-coronally and mesio-distally. Mucograft material will be prepared according to the manufacturer's instruction and trimmed as the size measured from the recipient and be placed and secured on the recipient bed with sutures.
  Interventions: Procedure: apically positioned flap with Mucograft

INTERVENTIONS:
Procedure: Apically positioned flap — Standard TUSDM Periodontology Clinic procedures will be followed. Local anesthesia will be achieved. Center of implant fixtures will be located. Crestal incision thru the center of implant fixture will be made. Implant fixture will be uncovered and healing abutment/s will be inserted. Horizontal incision at approximately 0.5mm coronal to buccalmucogingival junction will be made 1 tooth mesial to 1 tooth distal to the treating area.
  No vertical incision will be made Gingiva coronal to horizontal incision will remain intact Partial thickness flap will be prepared and displaced apically approximately 7mm from the horizontal incision and secured with sutures.
  Prepared surgical area will be measured apico-coronally and mesio-distally.
  Arms: Apically positioned flap
Procedure: Free Gingival Graft — Standard Clinic procedures followed. Local anesthesia achieved. Center of implant fixtures located. Crestal incision thru center of fixture will be made.
  Implant fixture uncovered and healing abutment/s inserted. Horizontal incision at approx 0.5mm coronal to buccalmucogingival junction will be made 1 tooth mesial to 1 tooth distal to the treating area.
  No vertical incision made. Gingiva coronal to horizontal incision remains intact.
  Partial thickness flap prepared and displaced apically approximately 7mm from horizontal incision; secured with sutures. Prepared recipient bed measured apico-coronally and mesio-distally. Masticatory mucosa from palate of treating side (Right or Left) harvested according to size measured from recipient bed with width of approximately 5mm at line of measurement. Harvested graft material will be transplanted on recipient bed, lined with initial horizontal incision line with sutures
  Arms: Free Gingival Graft
Procedure: apically positioned flap with Mucograft — Standard TUSDM Periodontology Clinic procedures followed. Local anesthesia achieved.
  Center of implant fixtures will be located. Crestal incision thru the center of implant fixture will be made. Implant fixture will be uncovered and healing abutment/s will be inserted. Horizontal incision at approximately 0.5mm coronal to buccalmucogingival junction will be made 1 tooth mesial to 1 tooth distal to the treating area.
  No vertical incision will be made. Gingiva coronal to horizontal incision will remain intact. Partial thickness flap will be prepared and displaced apically approximately 7mm from the horizontal incision and secured with sutures.
  Prepared recipient bed will be measured apico-coronally and mesio-distally. Mucograft material will be prepared according to the manufacturer's instruction and trimmed as the size measured from the recipient and be placed and secured on the recipient bed with sutures.
  Arms: Apically positioned flap with Mucograft

SUMMARY:
This research study is looking at three different procedures for improving the oral mucosa (membrane) around dental implants. The three procedures will be the standard procedure, the standard procedure with the use of tissue harvested from the mouth and the standard procedure with the use of Mucograft membrane product. An advantage claimed by the Mucograft manufacturer is increased patient comfort due to lack of tissue harvesting from the mouth. Pain and discomfort levels will be evaluated for each of the procedures. Gain in oral mucosa and the visual will also be evaluated.

DETAILED DESCRIPTION:
Experimental Design

The study design for this research project will be a single centered, prospective randomized controlled trial. Subjects will be Tufts University School of Dental Medicine Department of Periodontology patients.

Sample Size and Statistical Analysis

There will be up to 22 subjects in each group, with a total of up to 66 subjects in the study. Up to 80 subjects will be enrolled in order to have 66 subjects completed the study. The calculation is based on 2 point difference in VAS pain and discomfort survey to have 80% power, while setting α=0.025 to adjust for the two primary outcomes (pain and discomfort) which gives 19 per each group. However, considering a 15% drop out rate, up to 22 subjects for each group will be recruited.

Data collected for analysis will be 10 point VAS from subjects' survey forms for the primary outcome. And 10 point VAS from esthetic evaluation, gain of keratinized mucosa measured by periodontal probe in millimeters with stent will be data for secondary outcome.

For all variables, normality will be assessed using the Kolmogorov-Smirnov test. If the assumptions of normality hold, then means and standard deviations will be reported and the relationship between treatment arm and the outcome will be tested using one-way ANOVA. If the assumptions of normality do not hold, then medians and interquartile ranges will be reported and relationships will be tested using the Kruskal-Wallis test. If the initial analyses are significant, then the post hoc pair wise comparisons will be made using either independent sample t-tests or Mann-Whitney U-tests. When patients are lost to follow-up, their information will be excluded from the analyses. To account for the multiple comparisons, the Bonferroni correction will be implemented. Thus, all p-values less than 0.025 will be considered statistically significant. Analyses will be performed using SAS, Version 9.2 (SAS Institute, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for 2nd stage implant surgery at the periodontology clinic of TUSDM.
* Inadequate keratinized tissue (0.1mm- <2mm of buccal keratinized mucosa prior to the time of 2nd stage surgery) at the implant site. [4]
* Adequate depth of buccal vestibule (>7 mm from the crest of ridge, measured at the center of surgical area) to accommodate gain of keratinized mucosa width.

Exclusion Criteria:

* Lack of keratinized mucosa on the area of implant.
* Autoimmune conditions which may interfere with soft tissue healing in oral cavity, e.g., pemphigus vulgaris, phemphigoid
* Infectious disease (self-reported - HIV, tuberculosis or hepatitis)
* Pregnant patients, as part of TUSDM standard of care not to treat for non-emergency surgical procedures
* Uncontrolled diabetes, defined as HbA1c >=7, values measured within six months
* Previous gingival grafting procedure on the area.
* Smoking (>3 cigarettes per day)
* Subjects with known hypersensitivity to study materials or objection to use of porcine material (religious or cultural reasons)
* Known allergy to codeine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pain and discomfort survey | 10 to 14 days follow up
  A survey using VAS scale will be performed from the subjects at 10-14 days follow up visit.

SECONDARY OUTCOMES:
Evaluation of full mouth gingival condition (periodontal parameters) | At 3-month and 6-month follow up appointments.
  Subject's full mouth gingival condition will be evaluated using a periodontal probe. The following will be assessed at 4 sites/tooth: Plaque index (Modified O'Leary Plaque Index) and gingival index (Löe and Silness 1963). The following will be assessed at 6 sites/tooth: Probing depth (mm), Bleeding on probing (yes/no), Recession (mm), and Clinical attachment level (mm). Mobility (Miller classification) and mucogingival deformities will also be evaluated. Plaque control with oral hygiene instruction will be reinforced.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States